CLINICAL TRIAL: NCT06247098
Title: Sinus Augmentation Healing With Autogenous and Xenograft Mix Compared to Xenograft Alone
Brief Title: Evaluation of Sinus Augmentation Bone Healing Using Autograft and Xenograft Compared to Xenograft Alone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004629
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Sinus Floor Augmentation; Dental Implant; Bone Substitute; Autogenous Bone Graft
Keywords: Histology; Volume measurements; Radiographic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical examiners, study surgeons, and subjects will not be blinded. Analysis of histomorphometric, histologic, and volumetric data will be completed by an external lab and will not be aware of what group the subjects were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Xenograft - Autogenous 1:4 (Experimental): Sinus grafted with a ratio of Xenograft - Autogenous 1:4
  Interventions: Procedure: Sinus Lift augmentation; Device: Cone-beam computed tomography systems (CBCT)
- Xenograft alone (Active Comparator): Sinus grafted with Xenograft only
  Interventions: Procedure: Sinus Lift augmentation; Device: Cone-beam computed tomography systems (CBCT)

INTERVENTIONS:
Procedure: Sinus Lift augmentation — Randomised Sinus Lift augmentation either with Xenograft - Autogenous ratio 1:4 (test) or Xenograft alone (Control)
Device: Cone-beam computed tomography systems (CBCT) — An research only use of CBCT at visit 2 to review healing status.

SUMMARY:
To evaluate bone healing at 4 months after lateral sinus augmentation with a 4:1 ratio of autologous bone and xenograft or xenograft alone. A radiographic volumetric, histomorphometric, and histologic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Tufts School of Dental Medicine (TUSDM)
* Two stage sinus augmentations with <5mm (Zinner, Small 2004) residual bone height in need of augmentation for implant placement
* Full maxillary edentulism or Kennedy class I or III
* 18 to 100 year old

Exclusion Criteria:

* Adults unable to consent (cognitively impaired adults)
* Those who self-report as pregnant or breastfeeding
* Wards of the state
* Non-Viable neonates
* Neonates of uncertain viability
* < 18 years of age
* Refusal to participate
* Prior medical condition causing complications in bone metabolism
* Osteoporosis
* History of/or current chemotherapy
* History of/or current head and neck radiation
* Current heavy smoking > 10 cigarettes/day
* Self-reported pregnancy or lactation
* Previous history of sinus elevation procedure
* Existing sinus pathology or pathology discovered at time of sinus augmentation or implant placement
* Absence of autogenous donor site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Histological analysis | 4 months from surgery
  Mineralized and non-mineralized tissue Remnant particles of biomaterial Inflammatory infiltrate

SECONDARY OUTCOMES:
Volumetric bone analysis 4 months post sinus augmentation | 4 months from surgery
  Sinus volume calculation via CBCT analysis
Radiographic bone height gain at 4 months | 4 months post sinus augmentation
  Residual alveolar crest Final alveolar crest height at 4 months Initial height of graft immediately post graft placement Vertical bone material resorption

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Mordini, DDS, MS, Principal Investigator — Tufts Univeristy
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Moraissi E, Alhajj WA, Al-Qadhi G, Christidis N. Bone Graft Osseous Changes After Maxillary Sinus Floor Augmentation: A Systematic Review. J Oral Implantol. 2022 Oct 1;48(5):464-471. doi: 10.1563/aaid-joi-D-21-00310. PMID 35881815
- [Background] Al-Moraissi EA, Alkhutari AS, Abotaleb B, Altairi NH, Del Fabbro M. Do osteoconductive bone substitutes result in similar bone regeneration for maxillary sinus augmentation when compared to osteogenic and osteoinductive bone grafts? A systematic review and frequentist network meta-analysis. Int J Oral Maxillofac Surg. 2020 Jan;49(1):107-120. doi: 10.1016/j.ijom.2019.05.004. Epub 2019 Jun 21. PMID 31230768
- [Background] Barone A, Crespi R, Aldini NN, Fini M, Giardino R, Covani U. Maxillary sinus augmentation: histologic and histomorphometric analysis. Int J Oral Maxillofac Implants. 2005 Jul-Aug;20(4):519-25. PMID 16161735